CLINICAL TRIAL: NCT01913080
Title: The Use of a Health Management Tool in a Clinic Setting to Improve Self-Efficacy in Rheumatoid Arthritis Patients: a Randomized Clinical Trial.
Brief Title: The Health Log: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Nancy Shadick, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2013P000973
Record Dates: First submitted 2013-07-30; First posted 2013-07-31 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Rheumatoid Arthritis
Keywords: health management
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health Log (Active Comparator): Patients who have a billing diagnosis RA (714.0)or seronegative inflammatory arthritis who are enrolled in the Brigham and Women's Rheumatoid Arthritis Sequential Study (BRASS)will be given the Health Log health management tool.
  Interventions: Other: Health Log
- Control Pill Box (No Intervention): Controls will be BRASS patients who continue to receive regular care and are also given a pill box instead of the Health Log health management tool.

INTERVENTIONS:
Other: Health Log — The Health Log consists of a permanent booklet and a refillable health log version that is filled out before each doctor's appointment. The permanent booklet has areas to record:
  * Personal information and emergency contact(s)
  * Physician names and contact information
  * Insurance information
  * Medications, vitamins and supplements
  * Surgeries
  * Health history The booklet also includes suggested questions you may want to ask your Rheumatologist about medications, lifestyle, or future/status.
  The refillable health log includes questions about pain, fatigue,overall status from the Multi-Dimensional Health Assessment Questionnaire (MDHAQ), and a modified Arthritic Pain and Joint Evaluation. It also has space to write questions for the doctor's visit and prescription refills needed.
  Arms: Health Log

SUMMARY:
The goal of the present study is to determine if a health management tool improves self-efficacy, satisfaction with the doctor's visit, and agreement of the statement "How satisfied are you that your concerns were addressed during your clinic visit today" over time.

DETAILED DESCRIPTION:
The Patient-Centered Outcomes Initiative (PACO) was developed at Brigham and Women's Hospital (BWH) to create a replicable model of patient-centered care that will improve treatment for patients with rheumatoid arthritis (RA) and lead to improved outcomes. This work began with focus groups of RA patients to determine which changes or programs they felt were needed. Among the suggestions was a health management tool to improve doctor-patient communication. The Patient Advisory Committee (PAC), a part of PACO which grew out of the focus groups, worked to develop the current Health Log. It consists of a permanent booklet and a refillable health log version that is filled out before each doctor's appointment.

Health management tools have also been developed for patients with other chronic conditions. Dr. Paul Fortin of the University Health Network developed the Lupus Health Passport, which helps patients keep track of their health and also has information about lupus as well as prevention of coronary artery disease (CAD) and osteoporosis.

However, although these health management tools have been well received, they have not been studied to see if they improve self-efficacy. We would like to determine if the use of the Health Log improves self-efficacy in RA patients over time.

Specifically we will be looking to:

1. Determine if this health management tool improves self-efficacy over time with use, as measured by the Self-Efficacy Other Symptoms Scale of the Arthritis Self-Efficacy Questionnaire.
2. Determine if this health management tool improves satisfaction with the doctor's visit as measured by a VAS scale 10-100.
3. Determine if this health management tool improves agreement with the statement "How satisfied are you that your concerns were addressed during your clinic visit today", as measured by a VAS scale 10-100.

ELIGIBILITY:
Inclusion Criteria:

* billing diagnosis of rheumatoid arthritis (714.0) or seronegative inflammatory arthritis and a member of the BRASS study at Brigham and Women's Hospital

Exclusion Criteria:

* less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in Self-Efficacy | baseline and 12 months
  assessed using the Arthritis Self-Efficacy Scale

SECONDARY OUTCOMES:
Change in satisfaction with the doctor's visit | baseline and 12 months
  assessed using the VAS scale 10-100
Change in the statement "How satisfied are you that your concerns were addressed during your clinic visit today" | baseline and 12 months
  assessed using the VAS scale 10-100

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Shadick, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Linos A, Worthington JW, O'Fallon WM, Kurland LT. The epidemiology of rheumatoid arthritis in Rochester, Minnesota: a study of incidence, prevalence, and mortality. Am J Epidemiol. 1980 Jan;111(1):87-98. doi: 10.1093/oxfordjournals.aje.a112878. PMID 7352462
- [Background] Harris, E.D., Rheumatoid arthritis. 1997, Philadelphia: Saunders. xxiii, 433.
- [Background] Pincus T, Callahan LF, Sale WG, Brooks AL, Payne LE, Vaughn WK. Severe functional declines, work disability, and increased mortality in seventy-five rheumatoid arthritis patients studied over nine years. Arthritis Rheum. 1984 Aug;27(8):864-72. doi: 10.1002/art.1780270805. PMID 6431998
- [Background] Sherrer YS, Bloch DA, Mitchell DM, Young DY, Fries JF. The development of disability in rheumatoid arthritis. Arthritis Rheum. 1986 Apr;29(4):494-500. doi: 10.1002/art.1780290406. PMID 3707627
- [Background] Callahan LF, Brooks RH, Summey JA, Pincus T. Quantitative pain assessment for routine care of rheumatoid arthritis patients, using a pain scale based on activities of daily living and a visual analog pain scale. Arthritis Rheum. 1987 Jun;30(6):630-6. doi: 10.1002/art.1780300605. PMID 3606681
- [Background] Yelin E, Meenan R, Nevitt M, Epstein W. Work disability in rheumatoid arthritis: effects of disease, social, and work factors. Ann Intern Med. 1980 Oct;93(4):551-6. doi: 10.7326/0003-4819-93-4-551. PMID 7436187
- [Background] Meenan RF, Yelin EH, Henke CJ, Curtis DL, Epstein WV. The costs of rheumatoid arthritis. A patient-oriented study of chronic disease costs. Arthritis Rheum. 1978 Sep-Oct;21(7):827-33. doi: 10.1002/art.1780210714. PMID 100122
- [Background] Pincus T, Brooks RH, Callahan LF. Prediction of long-term mortality in patients with rheumatoid arthritis according to simple questionnaire and joint count measures. Ann Intern Med. 1994 Jan 1;120(1):26-34. doi: 10.7326/0003-4819-120-1-199401010-00005. PMID 8250453
- [Background] Lorig K, Chastain RL, Ung E, Shoor S, Holman HR. Development and evaluation of a scale to measure perceived self-efficacy in people with arthritis. Arthritis Rheum. 1989 Jan;32(1):37-44. doi: 10.1002/anr.1780320107. PMID 2912463
- [Background] Ware JE, Kosinski M, Keller SD. SF-12: How to Score the SF-12 Physical and Mental Health Summary Scales. 2nd ed. Boston, MA: The Health Institute, New England Medical Center; 1995.
- [Background] Wolfe F, Michaud K, Pincus T. Development and validation of the health assessment questionnaire II: a revised version of the health assessment questionnaire. Arthritis Rheum. 2004 Oct;50(10):3296-305. doi: 10.1002/art.20549. PMID 15476213
- [Background] Prevoo ML, van 't Hof MA, Kuper HH, van Leeuwen MA, van de Putte LB, van Riel PL. Modified disease activity scores that include twenty-eight-joint counts. Development and validation in a prospective longitudinal study of patients with rheumatoid arthritis. Arthritis Rheum. 1995 Jan;38(1):44-8. doi: 10.1002/art.1780380107. PMID 7818570
- See also: Website for the Health Log — http://www.pacostudy.org/tools-for-patients-and-doctors/